CLINICAL TRIAL: NCT02346331
Title: Epidemiology, Acute Management, and Outcomes of Patients With Sepsis Presenting to a Referral Hospital in Western Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Moi University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00056846; R25TW009337 (NIH)
Record Dates: First submitted 2015-01-14; First posted 2015-01-27 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WHO intervention (Experimental): This arm will be treated with the 2011 WHO sepsis recommendations for the first 6 hours of their hospitalization. The WHO recommendations involve fluid boluses guided by vital signs and physical exam, frequent patient monitoring, rapid and early administration of empiric antibiotics, oxygen delivery, correction of hypoglycemia, and correction of severe anemia.
  Interventions: Other: WHO algorithm of fluid boluses guided by physical examination; Other: Frequent patient monitoring; Other: Early administration of empiric antibiotics; Other: Oxygen delivery; Other: Correction of hypoglycemia; Other: Correction of severe anemia
- Standard care (No Intervention): This arm will be managed per standard care by the hospital clinicians.

INTERVENTIONS:
Other: WHO algorithm of fluid boluses guided by physical examination
  Arms: WHO intervention
Other: Frequent patient monitoring — Vital signs and physical exam every 30-60 minutes
  Arms: WHO intervention
Other: Early administration of empiric antibiotics — Clinician will be prompted to administer antibiotics within 60 minutes
  Arms: WHO intervention
Other: Oxygen delivery
  Arms: WHO intervention
Other: Correction of hypoglycemia — If blood glucose is less than 3.0 mmol/L, IV dextrose will be administered
  Arms: WHO intervention
Other: Correction of severe anemia — If hemoglobin is less than 7 mg/dL, clinician will be prompted to offer blood transfusion
  Arms: WHO intervention

SUMMARY:
Sepsis is a clinical syndrome representing deranged hemodynamics (such as tachycardia) secondary to severe infection. In high-income countries (HICs), early resuscitation of septic patients with protocol-driven therapy, including quantitative fluid administration guided by invasive monitoring, has resulted in improved outcomes for septic patients. Prevalence and mortality of sepsis are thought to be higher in sub-Saharan Africa (SSA) than in high-income countries; however, most hospitals in SSA lack the technology and resources necessary to implement the resuscitation protocols used in HICs and therefore, mortality from sepsis remains high. The World Health Organization (WHO) has recently disseminated an algorithm for resuscitation of septic patients in low resource settings. This algorithm is based on expert consensus only, and its efficacy has never been tested.

This study will be conducted in the Casualty Department of Moi Teaching and Referral Hospital (MTRH) in Eldoret, Kenya.

The purpose of this study is to describe the epidemiology of patients presenting with severe sepsis, to examine the microbiology causing severe sepsis, to describe current management and outcomes for severe sepsis, and to test the effect of implementation of the WHO resuscitation algorithm at MTRH.

The study design is a prospective before and after clinical trial. In an initial observational phase, adult patients presenting to the MTRH Casualty Department with sepsis and severe sepsis (the latter of which will be defined by elevated lactate) will be enrolled into a prospective observational cohort. Demographic data, medical characteristics, and microbiological studies will be obtained, then the management and outcomes of these patients will be observed. In a second phase, patients with sepsis will continue to be enrolled into a prospective observational cohort, while patients with severe sepsis will be enrolled into an intervention group. Patients in the intervention group will be managed according to the WHO resuscitation algorithm. Specifically, the WHO algorithm involves fluid boluses guided by vital signs and physical exam findings, rapid and early administration of empiric antibiotics, and frequent patient monitoring. The outcomes of interest are achievement of lactate clearance, which is a correlate of tissue perfusion, as well as 24-hour, in-hospital, and 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to MTRH Casualty Department for acute medical care
* Suspected infection, in the judgment of the managing clinician
* At least 2 of the following: axillary temperature >37.5°C or <35.5°C or core temperature >38.0°C or <36.0°C; heart rate >90 beats per minute; respiratory rate >20 breaths per minute; or systolic blood pressure <100 mmHg

Exclusion Criteria:

* Lack of basic language skills in either English or Kiswahili
* Pregnancy
* Congestive heart failure or valvular heart disease (as a known prior diagnosis or in the judgment of the managing clinician)
* Need for immediate surgery (within 6 hours) in the judgment of the managing clinician
* Inability to consent to study participation and lack of accompaniment by a family member or other surrogate who can provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Lactate clearance (difference in lactate [mmol/L] at study enrollment and 6 hours after study enrollment) as a measure of efficacy | enrollment, 6 hours
  Lactate level will be measured at study enrollment (time 0) and 6 hours after study enrollment (time 6). Lactate clearance will be reported as the difference between time 0 and time 6 lactate, as a fraction of time 0 lactate.

SECONDARY OUTCOMES:
Mortality | 24 hours, in-hospital, and 30 days
Number of subjects with adverse effects as a measure of safety | 6 hours, 24 hours, in-hospital, and 30 days

OTHER OUTCOMES:
Time of first antibiotic delivery | 1 hour
IV fluid volume (ml) | 6 hours, 24 hours, in-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Nathan M Thielman, MD, MPH, Principal Investigator — Duke University; Charles Kwobah, MBChB, MMed, Principal Investigator — Moi University
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Kenya